CLINICAL TRIAL: NCT04941079
Title: Safety and Efficacy of Inactivated SARS-CoV-2 Vaccine in Immune-related Myopathy (Myasthenia Gravis and Inflammatory Myopathy) Patients ：a Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Fei Xiao, Prof.Fei Xiao, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2021-296
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Myopathy
MeSH Terms: conditions — COVID-19; Muscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune-related Myopathy Patient (myasthenia gravis and inflammatory myopathy)
  Interventions: Other: no intervention
- Health Control
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study is a prospective observational study. We aim to investigate the safety and efficacy of inactivated SARS-CoV-2 vaccine between immune-related myopathy (myasthenia gravis and inflammatory myopathy) patients and health controls. The main study factors include adverse events following immunization (AEFI), serum specific antibody (Acetylcholine receptor (AChR) antibody, Anti-MuSK (muscle-specific kinase) antibody, myositis antibody) and virus neutralizing antibody titers.

ELIGIBILITY:
Inclusion Criteria:

1. Complete behavioral ability
2. Voluntary willingness to vaccinate
3. Clinically confirmed immune-related myopathy (myasthenia gravis and inflammatory myopathy) and immune-related myopathy (myasthenia gravis and inflammatory myopathy)was stable
4. Informed consent to the research

Exclusion Criteria:

1. No independent behavior ability
2. Vaccination is contraindicated
3. Other diseases that significantly affect the immune function
4. Other diseases that may significantly affect immune function are being treated
5. Vaccination contraindication was found during the study observation period
6. Other diseases that may significantly affect immune function were diagnosed during the study observation period
7. Treatments for other diseases that may significantly affect immune function were initiated during the study observation period
8. Refused regular follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Immune-related myopathy (myasthenia gravis and inflammatory myopathy) patients and health controls who are willing to receive two dose of SARS-CoV-2 inactivated vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events following immunization (AEFI) | 6 months
  Adverse event following immunization refers to any untoward medical occurrence which follows immunization and which does not necessarily have a causal relationship with the usage of the vaccine.
Serum specific antibody | 6 months
  Serum specific antibody of immune-related myopathy including Acetylcholine receptor (AChR) antibody, Anti-MuSK (muscle-specific kinase) antibody, myositis antibody.
Virus neutralizing antibody titer | 6 months
  Virus neutralizing antibody titer of Covid-19.

IPD SHARING:
Plan to Share IPD: Undecided
Undeicded